CLINICAL TRIAL: NCT06111573
Title: Comparative Evaluation of the Effectiveness of Diclofenac Sodium Versus Vitamin D Supplements on Symptoms in Individuals With Myofascial Pain and Vitamin D Deficiency
Brief Title: Comparative Evaluation of the Effectiveness of Diclofenac Sodium Versus Vitamin D on Myofascial Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Serap Keskin Tunc, Associate Professor, Yuzuncu Yil University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: YYU-10/31.05.2023
Record Dates: First submitted 2023-10-26; First posted 2023-11-01 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Myofascial Pain Dysfunction Syndrome,Temporomandibular Joint
Keywords: temporomandibular joint; vitamin d; myofascial pain; sodium diclofenac
MeSH Terms: conditions — Temporomandibular Joint Dysfunction Syndrome | interventions — Vitamin D; Diclofenac

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin D + Occlusal Splint (Experimental): Vitamin D is a fat-soluble secosteroid. Vitamin D is very important in muscle and bone metabolism. Vitamin D is a vitamin with some anti-inflammatory and immune-modulating properties.
  Interventions: Dietary Supplement: Vitamin D
- Diclofenac Sodium + Occlusal Splint (Active Comparator): Diclofenac Sodium is a type of NSAID which has been found effective both as an analgesic and in reducing inflammation and is classified as weak and preferentially COX-2 selective.
  Interventions: Drug: Diclofenac Sodium

INTERVENTIONS:
Dietary Supplement: Vitamin D — Study group using Vitamin D for myofascial pain treatment. "Diagnostic Criteria for Temporomandibular Disorders" was used in the diagnosis of patients with myofascial pain. Study group usind Vitamin D for myofascial pain treatment. Medical treatment with Vitamin D (10,000 IU/day) + Occlusal Splint treatment was applied. Occlusal Splints were made of hard acrylic with a flat surface and were used only for 8 hours during sleep for 3 months. 500 mg Paracetamol tablet was prescribed to the patients as a rescue painkiller if they needed painkillers.
  Other Names: devit-3
  Arms: Vitamin D + Occlusal Splint
Drug: Diclofenac Sodium — "Diagnostic Criteria for Temporomandibular Disorders" was used in the diagnosis of patients with myofascial pain. Control group using Diclofenac Sodium for myofascial pain treatment. Medical treatment with Diclofenac Sodium (Voltaren 75 mg, 2x1 ) + Occlusal Splint treatment was applied. Occlusal Splints were made of hard acrylic with a flat surface and were used only for 8 hours during sleep for 3 months. 500 mg Paracetamol tablet was prescribed to the patients as a rescue painkiller if they needed painkillers.
  Other Names: Voltaren
  Arms: Diclofenac Sodium + Occlusal Splint

SUMMARY:
It has been reported in the literature that there is a significant relationship between bruxism and low serum vitamin D levels. It was aimed to compare the effectiveness of diclofenac sodium treatment versus vitamin D supplementation on symptoms in individuals with myofascial pain and vitamin D deficiency.

DETAILED DESCRIPTION:
In the current literature, it has been reported that there is a significant relationship between teeth grinding and low serum vitamin D levels. Vitamin D has been shown to play an important role in the musculoskeletal and cardiovascular systems, as well as in the control of calcium and phosphate metabolism and in maintaining adequate blood levels of these minerals. Vitamin D deficiency has been associated with poor physical performance and low muscle strength. There are also studies to understand the relationship between TMJ disorders and vitamin D level (serum 25(OH) D). These studies reported a relationship between the presence of TMJ disorder and vitamin D deficiency.

NSAIDs are a large group of drugs that inhibit cyclooxygenases and thus prevent the formation of prostaglandins. Traditionally, it has been the most commonly prescribed group of medications for pain in the orofacial area. It is recommended to use these drugs regularly for at least 2 weeks to achieve an anti-inflammatory effect in individuals with TMJ disorders.

It was aimed to compare the effectiveness of diclofenac sodium treatment versus vitamin D supplementation on symptoms in individuals with myofascial pain and vitamin D deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Vitamin D deficiency,
* Myofascial pain complaint,
* Chronic pain,
* No missing teeth,
* Absence of open bite and/or crossbite.

Exclusion Criteria:

* Individuals who have undergone interventional or surgical procedures related to the temporomandibular joint,
* Temporomandibular joint pathology,
* Pregnancy or breastfeeding,
* Individuals who do not come for postoperative checks,
* Using different medications other than those recommended,
* Allergy to study drugs and materials to be used

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
VAS pain score | At baseline
  A Visual Analogue Scale (VAS) is one of the pain rating scales between 1-10.
VAS pain score | 1 week
  A Visual Analogue Scale (VAS) is one of the pain rating scales between 1-10.
VAS pain score | 1 mounth
  A Visual Analogue Scale (VAS) is one of the pain rating scales between 1-10.
VAS pain score | 3 mounth
  A Visual Analogue Scale (VAS) is one of the pain rating scales between 1-10.
Painless Unassisted Mouth Opening | At baseline
  Pain-free opening e.g. maximum comfortable opening was defined as the maximum distance the subject could open his/her mouth without experiencing any pain and discomfort. After the subject had opened this wide, the examiner measured the distance between the maxillary and mandibular incisal edges.
Painless Unassisted Mouth Opening | 1 week
  Pain-free opening e.g. maximum comfortable opening was defined as the maximum distance the subject could open his/her mouth without experiencing any pain and discomfort. After the subject had opened this wide, the examiner measured the distance between the maxillary and mandibular incisal edges.
Painless Unassisted Mouth Opening | 1 mounth
  Pain-free opening e.g. maximum comfortable opening was defined as the maximum distance the subject could open his/her mouth without experiencing any pain and discomfort. After the subject had opened this wide, the examiner measured the distance between the maxillary and mandibular incisal edges.
Painless Unassisted Mouth Opening | 3 mounth
  Pain-free opening e.g. maximum comfortable opening was defined as the maximum distance the subject could open his/her mouth without experiencing any pain and discomfort. After the subject had opened this wide, the examiner measured the distance between the maxillary and mandibular incisal edges.
Maximum Unassisted Mouth Opening | At baseline
  Maximum assisted opening was defined as the maximum distance the subject could open the mouth, even if he/she felt pain or discomfort. The interincisal distance between the maxillary and mandibular incisal edges was measured.
Maximum Unassisted Mouth Opening | 1 week
  Maximum assisted opening was defined as the maximum distance the subject could open the mouth, even if he/she felt pain or discomfort. The interincisal distance between the maxillary and mandibular incisal edges was measured.
Maximum Unassisted Mouth Opening | 1 mounth
  Maximum assisted opening was defined as the maximum distance the subject could open the mouth, even if he/she felt pain or discomfort. The interincisal distance between the maxillary and mandibular incisal edges was measured.
Maximum Unassisted Mouth Opening | 3 mounth
  Maximum assisted opening was defined as the maximum distance the subject could open the mouth, even if he/she felt pain or discomfort. The interincisal distance between the maxillary and mandibular incisal edges was measured.
Maximum Assisted Mouth Opening | At baseline
  Maximum assisted opening was defined as the maximum distance the subject could open the mouth, even if he/she felt pain or discomfort. After the subject had opened this wide, the examiner placed his fingers on the subject's maxillary and mandibular central incisors, and forced the subject's mouth to open wider. The interincisal distance between the maxillary and mandibular incisal edges was measured.
Maximum Assisted Mouth Opening | 1 week
  Maximum assisted opening was defined as the maximum distance the subject could open the mouth, even if he/she felt pain or discomfort. After the subject had opened this wide, the examiner placed his fingers on the subject's maxillary and mandibular central incisors, and forced the subject's mouth to open wider. The interincisal distance between the maxillary and mandibular incisal edges was measured.
Maximum Assisted Mouth Opening | 1 mounth
  Maximum assisted opening was defined as the maximum distance the subject could open the mouth, even if he/she felt pain or discomfort. After the subject had opened this wide, the examiner placed his fingers on the subject's maxillary and mandibular central incisors, and forced the subject's mouth to open wider. The interincisal distance between the maxillary and mandibular incisal edges was measured.
Maximum Assisted Mouth Opening | 3 mounth
  Maximum assisted opening was defined as the maximum distance the subject could open the mouth, even if he/she felt pain or discomfort. After the subject had opened this wide, the examiner placed his fingers on the subject's maxillary and mandibular central incisors, and forced the subject's mouth to open wider. The interincisal distance between the maxillary and mandibular incisal edges was measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Van Yüzüncü Yıl University, Van, Turkey (Türkiye)

REFERENCES:
- [Derived] Kahraman NH, Tunc SK. Comparative evaluation of the effects of diclofenac sodium and vitamin D supplementation on symptoms in individuals with myofascial pain and vitamin D deficiency: a randomized controlled clinical trial. BMC Oral Health. 2025 Aug 29;25(1):1383. doi: 10.1186/s12903-025-06729-1. PMID 40883693